CLINICAL TRIAL: NCT05284695
Title: CAN POSTOPERATIVE PAIN BE PREVENTED in BARIATRIC SURGERY? EFFICACY and USABILITY of FASCIAL PLANE BLOCKS: a RETROSPECTIVE CLINICAL STUDY
Brief Title: The EFFICIENCY of FASCIAL PLANE BLOCKS in BARIATRIC SURGERY
Status: Completed | Type: Observational
Sponsor: V.K.V. American Hospital, Istanbul (Other)
Responsible Party: Principal Investigator, Sami Kaan Coşarcan, MD, V.K.V. American Hospital, Istanbul
Other Study IDs: Cosarcan4
Record Dates: First submitted 2022-02-25; First posted 2022-03-17 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2022-03

CONDITIONS: Regional Anesthesia Morbidity; Post Operative Pain; Bariatric Surgery Candidate
MeSH Terms: conditions — Pain, Postoperative | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- TAP + RB: transversus abdominis plane block and rectus sheath block
  Interventions: Procedure: Bariatric surgery
- ESPB: Erector spinae plane block
  Interventions: Procedure: Bariatric surgery
- EOI: External oblique intercostal block
  Interventions: Procedure: Bariatric surgery

INTERVENTIONS:
Procedure: Bariatric surgery — Patients undergoing elective bariatric surgery

SUMMARY:
Bariatric surgery effectively produces weight loss and reduces obesity-related comorbidities. Although it is mostly performed with minimally invasive techniques, the patients may still suffer from moderate-to-severe pain immediately after surgery [1]. Opioids remain the first choice for multimodal analgesia in the treatment of postoperative pain. Providing analgesia after bariatric surgery might be challenging due to a high prevalence of obstructive sleep apnea syndrome and the increased sensitivity to respiratory depression triggered by opioid overuse after surgeryThe most common plane block techniques utilized during laparoscopic bariatric surgery are transversus abdominis plane block (TAP), rectus sheath block (RB), the erector spinae plane block (ESPB) and the external oblique intercostal block (EOI). In this study, we have evaluated the auxiliary benefit of these various techniques in reduction of the postoperative in bariatric surgery. patients who had laparoscopic bariatric surgery at VKV American Hospital between January 2019 and December 2021 were reviewed retrospectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective bariatric surgery

Exclusion Criteria:

* Patients with a history of cerebrovascular events
* Alzheimer's and dementia
* inadequate cognitive functions
* history of chronic pain
* long-term opioid therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Fascial plane blocks and postoperative analgesia efficacy were investigated in bariatric surgery patients.
Sampling Method: Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
postoperative analgesia | 0 - 24 hours
  Postoperative pain assessment of patients will be made with a numeric rating scale (NRS). Postoperative opioid consumption will be examined

CONTACTS AND LOCATIONS:
Overall Officials: sami kaan coşarcan, Study Chair — American hospital
Locations (1):
- American Hsopital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Park CH, Nam SJ, Choi HS, Kim KO, Kim DH, Kim JW, Sohn W, Yoon JH, Jung SH, Hyun YS, Lee HL; Korean Research Group for Endoscopic Management of Metabolic Disorder and Obesity. Comparative Efficacy of Bariatric Surgery in the Treatment of Morbid Obesity and Diabetes Mellitus: a Systematic Review and Network Meta-Analysis. Obes Surg. 2019 Jul;29(7):2180-2190. doi: 10.1007/s11695-019-03831-6. PMID 31037599
- [Background] Subramani Y, Nagappa M, Wong J, Patra J, Chung F. Death or near-death in patients with obstructive sleep apnoea: a compendium of case reports of critical complications. Br J Anaesth. 2017 Nov 1;119(5):885-899. doi: 10.1093/bja/aex341. PMID 29077813
- [Background] Frauenknecht J, Kirkham KR, Jacot-Guillarmod A, Albrecht E. Analgesic impact of intra-operative opioids vs. opioid-free anaesthesia: a systematic review and meta-analysis. Anaesthesia. 2019 May;74(5):651-662. doi: 10.1111/anae.14582. Epub 2019 Feb 25. PMID 30802933
- [Background] Brummett CM, Waljee JF, Goesling J, Moser S, Lin P, Englesbe MJ, Bohnert ASB, Kheterpal S, Nallamothu BK. New Persistent Opioid Use After Minor and Major Surgical Procedures in US Adults. JAMA Surg. 2017 Jun 21;152(6):e170504. doi: 10.1001/jamasurg.2017.0504. Epub 2017 Jun 21. PMID 28403427
- [Background] Chin KJ, McDonnell JG, Carvalho B, Sharkey A, Pawa A, Gadsden J. Essentials of Our Current Understanding: Abdominal Wall Blocks. Reg Anesth Pain Med. 2017 Mar/Apr;42(2):133-183. doi: 10.1097/AAP.0000000000000545. PMID 28085788
- [Derived] Cosarcan SK, Yavuz Y, Dogan AT, Ercelen O. Can Postoperative Pain Be Prevented in Bariatric Surgery? Efficacy and Usability of Fascial Plane Blocks: a Retrospective Clinical Study. Obes Surg. 2022 Sep;32(9):2921-2929. doi: 10.1007/s11695-022-06184-9. Epub 2022 Jul 1. PMID 35776242